CLINICAL TRIAL: NCT02589756
Title: Fish or Nuts? Dietary Effects on Cardiometabolic Risk Factors and Persistent Organic Pollutants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Sasa Dusanov, PhD candidate, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015FO7650
Record Dates: First submitted 2015-09-14; First posted 2015-10-28 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Obesity; Metabolic Syndrome; Diabetes
Keywords: obesity; persistent organic pollutants; metabolic syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- The fatty fish group (Experimental): Participants will eat fatty fish and avoiding nuts)
  Interventions: Other: The nut group; Other: The control group
- The nut group (Experimental): Participants who will avoid fatty fish
  Interventions: Other: The fatty fish group; Other: The control group
- The control group (Placebo Comparator): Participants who will avoid both fatty fish and nuts
  Interventions: Other: The fatty fish group; Other: The nut group

INTERVENTIONS:
Other: The fatty fish group — At inclusion demographic information recorded, including length of breastfeeding for women. Thereafter, participants will start with a run-in period of two weeks where they will be asked not to consume salmon, mackerel, sardines or other fatty fish or nuts providing a dietary baseline. At baseline, subjects will be randomized to a fish, nuts or control group. The fish group will be asked to consume three to four portions weekly. The fish will be eaten at the main meal and in sandwiches for a total of 600 grams weekly for 6 months. This group will avoid eating nuts. The nut group will consume equal amount of energy (~1400 kcal ) for weekly use for 6 months. This group will avoid eating fatty fish. The control group will consume their usual diet, but asked to avoid fatty fish and nuts.
  Arms: The control group; The nut group
Other: The nut group — At baseline (conditions for baseline are the same in all three groups) the nut group will consume equal amount of energy (~1400 kcal ~100 grams walnuts, ~50 grams hazelnuts and ~50 grams almonds/week).The nuts will be provided free of charge for the six months. This group will avoid eating fatty fish.
  Arms: The control group; The fatty fish group
Other: The control group — After the baseline the control group will consume their usual diet, asked to avoid fatty fish and nuts.
  Arms: The fatty fish group; The nut group

SUMMARY:
Obesity represents one of the most important public health challenges for the societies. Although excess energy intake and physical inactivity are major causes of obesity and cardiometabolic disorders, emerging evidence has linked persistent organic pollutants (POPs) with the global epidemic of type 2 diabetes. However, the potential impacts of POPs on obesity and cardiometabolic risk in humans remain poorly known. On the other side systematic reviews and meta-analyses conducted in recent years strongly support a protective association between eating nuts and CVD. The investigators will conduct a randomized controlled clinical trial in adults. The main research questions are: a. Does consumption of fatty fish increase levels of POPs in overweight and obese adult norwegian men and women compared to a control group not consuming fatty fish? b. Does consumption of fatty fish affect markers of cardiometabolic risks (blood pressure, lipids, glucose and CRP) in overweight and obese adult norwegian men and women compared to a control group not consuming fatty fish? c. Does consumption of nuts improve markers of cardiometabolic risks in overweight and obese adult Norwegian men and women compared:1. to a control group not consuming nuts or fatty fish and 2. to a group consuming fatty fish.

Clinical significance of study: If an increase in POP levels is seen, and correlates with cardiometabolic risks, this may indicate the need to look further at a causal relation between POPs and cardiometabolic disease and risk factors particularly type 2 diabetes. If eating nuts improves CVD risk factors compared to not eating nuts, or to eating fatty fish, this could be important dietary information for populations at high risk of CVD.

DETAILED DESCRIPTION:
Today more than one-fifth of the adult Norwegian population is obese, and the prevalence of abdominal obesity has increased disproportionately in women. Cardiometabolic disorders (metabolic syndrome, type 2 diabetes) follow in the wake of obesity increasing health burdens on the population. Persistent organic pollutants (POPs) are lipophilic chemicals like dioxins, polychlorinated biphenyls (PCBs), and organochlorine pesticides (OPs) that bioaccumulate in living organisms for many years. In humans POPs are mainly stored in adipose tissue, and these chemicals have been detected in plasma of all populations, including babies. Humans are mainly exposed to POPs through the consumption of fatty rich food, with the highest levels of POPs being present in fatty fish. Because of the presence of polyunsaturated n-3 fatty acids, eating fatty fish has been generally associated with good health outcomes. However, questions have arisen whether POPs and other pollutants are impairing the nutritional benefits of fish (5). Dietary modification is a major cornerstone of prevention and treatment of obesity and cardiovascular disease (CVD). Evidence has linked the Mediterranean diet to prevention of CVD and sustained weight loss. The Mediterranean diet as consumed traditionally consists of bread, legumes, vegetables and fruits, nuts, olive oil, and limited red meats, meat products, butter, hard margarine and sugar as well as moderate alcohol intake. Acceptance and feasibility of the Mediterranean diet is limited in non-Mediterranean countries and in certain groups and requires modification according to local culture and norms. In Norway, official dietary recommendations advise that the population should eat lots of vegetables, fruit, berries, whole grains, legumes, nuts and fish and that processed and red meats, salt and sugar should be limited (11). Nuts are a powerhouse of protein, fiber, unsaturated fatty acids including n-3 fatty acids and phytochemicals, and are easy to incorporate into the diet. Evidence links nuts to reduced rates of CVD and overweight. Dietary recommendations most likely to reduce CVD risk in patients with overweight or obesity are controversial. If eating fatty fish regularly worsens metabolic regulation, an alternative to fatty fish may be eating nuts. This study aims to clarify the effects of eating fatty fish compared to nuts on cardiovascular risk factors and levels of POPs in patients with overweight or obesity who are at risk of CVD. 2.0 Insulin resistance is tightly related to abdominal obesity and is accompanied by a host of changes in cardiometabolic risk factors including low HDL cholesterol, high triglycerides, and subclinical inflammation (shown as high CRP), disturbances that lead to CVD. Other characteristics include high levels of adipokines (leptin, visfatin) and decreased adiponectin, an insulin-sensitizing hormone. Clinically the presence of three or more of five risk factors, namely abdominal obesity, low HDL cholesterol, high triglycerides, high fasting glucose, and high blood pressure, characterizes metabolic syndrome. Insulin resistance can be measured most precisely by the hyperinsulinemic euglycemic clamp method, but this method is time consuming and can only be applied to limited samples. Clinically, insulin resistance is suggested by high C-peptide. The Homeostasis Model Assessment index can be calculated to estimate insulin resistance (HOMA-IR) using fasting glucose and insulin levels. 3.1 Obesity and POPs Factors affecting the homeostasis between POPs stored in adipose tissue and circulating blood concentrations are not clear. Both higher and lower POP levels have been reported in obese versus lean individuals. These associations may differ according to the compound and previous exposure. Less chlorinated PCBs, dichlorodiphenyldichloroethylene (DDE) and dioxin showed adjusted odds ratio of 2-3 for abdominal obesity in data from seniors. Because studies are mostly cross-sectional, or obtained data on weight change retrospectively, causation between POP levels and obesity remains speculative. Weight loss reduces adipose tissue storage increasing concentrations in blood in the short term, though drastic weight loss decreases the total body burden. 3.3 Farmed fish as a source of POPs - studies from Norway A much cited study published in 2004 found that farmed salmon had significantly higher POP burdens than wild salmon and that farmed salmon from Europe were significantly more contaminated than farmed salmon from South and North America. Since that time, levels of some POPs like dioxins are likely to have decreased, as current aquaculture feed increasingly is based on plant oils. However, other contaminants like OPs and polycyclic aromatic hydrocarbons (PAH), which are omnipresent in vegetable oils, are largely present in farmed fish. Recently, significant amounts of POPs were reported to remain in Norwegian salmon. Importantly, proportions of n-3 fatty acids have decreased by about 50%. High levels of POPs have been shown in coastal Norwegian populations, as well as associations between marine food consumption and concentrations of POPs (26, 27). Further studies have shown that oily fish is the main source of PCBs and dioxins in both high and population-representative fish consumers in Norway. Clear correlations were shown between estimated intakes and blood concentrations of POPs. 4.1 Nuts and CVD Systematic reviews and meta-analyses conducted in recent years strongly support a protective association between eating nuts and CVD. Three meta-analyses appeared in 2014. Studies found that nut intake was inversely associated with ischemic heart disease, overall CVD and all-cause mortality but not significantly associated with diabetes and stroke. There was found an inverse association between eating nuts and incident ischemic heart disease and diabetes but not with stroke. It has been found a linear dose-response relationship between nut consumption and coronary artery disease (CAD) risk, where the risk of CAD decreased by 5% for every serving/week. Randomized dietary trial provided experimental evidence to support the protective effect of nuts on CVD. Participants aged 55 to 80 years and at high risk of CVD were randomly assigned to one of three dietary interventions: Mediterranean diet supplemented with virgin olive oil or nuts (approximately 30 g/day of mixed nuts), or a low-fat diet. The primary end point was the rate of major cardiovascular events (myocardial infarction, stroke, or death from cardiovascular causes) and median follow-up was 4.8 years. The multivariable-adjusted hazard ratio for the group assigned to a Mediterranean diet with nuts was 0.72 versus the control group. 4.2 Nuts and body weight Though nuts are an energy dense food, eating nuts does not appear to be associated with increased body weight. Meta-analysis conducted in 2013 found 33 relevant clinical trials of nut intake that provided outcomes of body weight. Compared with control diets, diets enriched with nuts did not increase body weight, BMI or waist circumference. The effects of nuts on energy have been summarized lately. Nuts are characterized as having high satiety value leading to strong compensatory dietary responses, inefficiency in absorption of the energy they contain and augmentation of fat oxidation. 4.3 Nuts and cardiometabolic risk factors A number of mechanisms have been examined in experimental studies providing putative explanations of the protective effects of nuts on CVD. Effects have been shown primarily with walnuts, hazelnuts, almonds and pistachios. Eating walnuts was shown to improved endothelial function in overweight adults with visceral obesity. Mediterranean diets supplemented with olive oil or nuts reduced 24-hour ambulatory blood pressure, total cholesterol and fasting glucose and reversed metabolic syndrome and shifted lipoprotein subfractions to a less atherogenic pattern. Diets enriched with hazelnuts improved endothelial function, prevented LDL oxidation and lowered inflammatory markers in addition to lipid-lowering effects. Nuts could be an alternative to fatty fish in the diet, both for persons wishing to eat vegetarian diets, for those wishing to avoid contaminants, and for improving CVD risk factors in persons at high risk. However, we are unaware of studies that have compared CVD risk factors in diets including nuts versus fatty fish.

5.0 Objectives of the study and main hypotheses

1. to a control group not consuming nuts or fatty fish
2. to a group consuming fatty fish

Hypotheses:

1. The investigators hypothesize that consumption of fatty fish will increase levels of POPs in overweight and obese norwegian men and women.
2. The investigators hypothesize that the consumption of fatty fish will change markers of cardiometabolic risk in overweight and obese norwegian men and women.
3. The investigators hypothesize that the consumption of nuts will improve markers of cardiometabolic risks in overweight and obese norwegian men and women both compared to a control group not consuming nuts and to the group consuming fatty fish. Variables, follow-up and endpoints: Clinic visits will be scheduled at biweekly intervals during the first 12 weeks to ensure stability of body weight in both groups and compliance. Vital signs and weight will be measured at visits in a standardized manner. A subsample of 15 participants in each of the fish, nut and control groups will undergo a hyperinsulinemic euglycemic clamp for evaluation of insulin sensitivity and resistance at baseline and after three months. For POPs analyses samples will be frozen at -70 degrees Celsius and analyzed batchwise for the following 21 POPs, which are suspected to strongly act as endocrine and metabolic disruptors:14 PCBs, including dioxin-like PCBs and non-dioxin-like PCBs, 5, 2,2',4,4'-tetra-bromobiphenyl ether and 1 dioxin. Power: Similar studies to the current one have not been performed previously to help in calculation of sample size, however, this is attempted. In a six-month period a possibly clinically relevant change in POPs may be a 15-20% increase - this is also the difference in PCBs between representative and high consumers in Norway (29). The study will include 40 participants in each group to allow for dropouts for a total of 120 participants. Clinical significance of study: If an increase in POP levels is seen, and correlates with cardiometabolic risks, this may indicate the need to look further at a causal relation between POPs and cardiometabolic disease and risk factors particularly type 2 diabetes. If eating fatty fish promotes cardiometabolic risk, this may indicate the need to reevaluate current dietary recommendations. If eating nuts improves CVD risk factors compared to not eating nuts, or to eating fatty fish, this could be important dietary information for populations at high risk of CVD.

4.3 Statistical analyses The statistical analysis will follow intent-to-treat principle, with additional complementary analyses of the per protocol population. Data analysis for changes in POPs and CVD risk factors will comprise all randomized individuals who complete the 12-week first study phase (intention to treat analysis - primary outcome). This analysis will be repeated including only per protocol participants who recorded over 80% compliance with assigned foods (completer analysis - secondary outcome). Between group comparisons of changes in POPs and CVD risk factors will be performed using the independent samples t-test. The study will compare the fish group to controls, and to the nut group. Within-group comparisons will be performed using the paired t-test. P-values <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40 to 65 years
* BMI in the overweight (25-29.9) or obese (30-34.9)
* Range and components of metabolic syndrome (waist circumference >102 cm for men or >94 cm for women; fasting glucose >5.6 mmol/l, HDL cholesterol <1.3 for women or <1.0 for men, and triglycerides >1.7 mmol/l)
* Fertile women are required to use reliable contraception

Exclusion Criteria:

* Cigarette smoking
* Diabetes mellitus
* Allergy or dislike of fish
* allergy or dislike of nuts
* chronic disease
* morbid obesity due to ethical reasons and weight fluctuations
* eating disorder

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
persistent organic pollutants | 6 months
  Measuring of persistent organic pollutants' levels before and after intervention.
  Blood tests will be obtained at randomization, and six months of follow-up for analysis analysis of environmental pollutants including 21 POPs in g/mol .Six-month follow-up samples will be stored for future analyses.

SECONDARY OUTCOMES:
waist circumference | 6 months
  waist circumference in cm as cardiometabolic risk factor
Parameter of inflammation CRP (C-reactive protein) | 6 months
  Secondary endpoints will include C-reactive protein
Parameter of insulin resistance HOMA index | 6 months
  The HOMA index (The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance and beta-cell function) in % will be calculated
C-peptide | 6 months
  C-peptide in nmol/L
Insulin | 6 months
  insulin in pmol/L
HbA1C | 6 months
  Hba1c in %
Glucose | 6 months
  fasting glucose in mmol/L
HDL-C | 6 months
  HDL-C (high-density lipoprotein) in mmol/L
Blood Pressure | 6 months
  Blood pressure in mm Hg
Triglycerides | 6 months
  Triglycerides in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Kare I Birkeland, MD, Ph.D, Study Director — Department of Endocrinology, Morbid Obesity and Preventive Medicine, Oslo University Hospital, Norway
Locations (1):
- Oslo University Hospital, Ullevål, Oslo, Norway

REFERENCES:
- [Background] Ngwa EN, Kengne AP, Tiedeu-Atogho B, Mofo-Mato EP, Sobngwi E. Persistent organic pollutants as risk factors for type 2 diabetes. Diabetol Metab Syndr. 2015 Apr 30;7:41. doi: 10.1186/s13098-015-0031-6. eCollection 2015. PMID 25987904
- [Background] Schecter A, Colacino J, Haffner D, Patel K, Opel M, Papke O, Birnbaum L. Perfluorinated compounds, polychlorinated biphenyls, and organochlorine pesticide contamination in composite food samples from Dallas, Texas, USA. Environ Health Perspect. 2010 Jun;118(6):796-802. doi: 10.1289/ehp.0901347. Epub 2010 Feb 10. PMID 20146964
- [Background] Tan SY, Dhillon J, Mattes RD. A review of the effects of nuts on appetite, food intake, metabolism, and body weight. Am J Clin Nutr. 2014 Jul;100 Suppl 1:412S-22S. doi: 10.3945/ajcn.113.071456. Epub 2014 Jun 11. PMID 24920033
- [Background] Orem A, Yucesan FB, Orem C, Akcan B, Kural BV, Alasalvar C, Shahidi F. Hazelnut-enriched diet improves cardiovascular risk biomarkers beyond a lipid-lowering effect in hypercholesterolemic subjects. J Clin Lipidol. 2013 Mar-Apr;7(2):123-31. doi: 10.1016/j.jacl.2012.10.005. Epub 2012 Oct 26. PMID 23415431
- [Derived] Dusanov S, Svendsen M, Ruzzin J, Kiviranta H, Gulseth HL, Klemsdal TO, Tonstad S. Effect of fatty fish or nut consumption on concentrations of persistent organic pollutants in overweight or obese men and women: A randomized controlled clinical trial. Nutr Metab Cardiovasc Dis. 2020 Mar 9;30(3):448-458. doi: 10.1016/j.numecd.2019.11.006. Epub 2019 Nov 21. PMID 32008913